# INFORMED CONSENT FORM AND

# **AUTHORIZATION TO USE AND DISCLOSE PROTECTED HEALTH INFORMATION**

Sponsor / Study Title: Melissa A Geller, MD - University of Minnesota /

"Intraperitoneal FT538 with Intravenous Enoblituzumab in Recurrent Ovarian, Fallopian Tube, and Primary Peritoneal

Cancer"

Protocol Number: CPRC # 2021LS103 (MT2021-27)

**Principal Investigator:** 

(Study Doctor)

Melissa Geller, MD

Telephone: 612-626-3111

612-273-3000 (24-Hour)

Address: University of Minnesota

420 Delaware St. SE Minneapolis, MN, 55455

If your doctor is Dr. Geller, please note that she is interested in both your medical care and the conduct of this research study. You have the right to discuss this study with another person who is not part of the research team before deciding whether to participate in the research.

**Supported By:** The research related expenses for this study are covered by National Institutes of Health (NIH) grants.

Fate Therapeutics is supplying the FT538 cell product without cost for the purpose of this study. MacroGenics, Inc. is supplying enoblituzumab without cost for the purpose of this study.

**Financial Interest Disclosure:** This research is supported in part by Fate Therapeutics. The University of Minnesota has licensed certain aspects of FT538, the cell product being tested in this study, to Fate Therapeutics. The University of Minnesota may benefit financially if the product is marketed in the future.

The University of Minnesota has a financial interest in the FT538 cell treatment due to its license agreement with Fate Therapeutics, which is providing the FT538 for this study. This interest has been reviewed and managed by the University of Minnesota in accordance with its conflict of interest policies. If you would like further information about this interest, please contact Jon Guden, Associate Director, Conflict of Interest Program, at jguden@umn.edu

### **Key Information About This Research Study**

The following is a short summary to help you decide whether or not to be a part of this research study. More detailed information is listed later in this form.

## What is research?

The study doctors are committed to your care and safety. There are important differences between research and treatment plans:

- The goal of research is to learn new things in order to help groups of people in the future. Study doctors learn things by following the same plan with a number of participants. You, as an individual, may or may not be helped by participating in a research study; however, your participation helps answer the research questions.
- The goal of routine (standard) treatment is to treat your cancer. Standard treatments are available from any doctor.

Research and clinical care are often combined. One purpose of this consent document is to provide you clear information about the specific research activities of this study. This consent form is to help you decide if you want to participate in the research study. You should not join this research study until all your questions are answered.

## Why am I being asked to take part in this research study?

You are invited to take part in this research study because you have ovarian, fallopian tube or primary peritoneal cancer that has returned (recurred) despite previous treatment.

## Things to Know Before Deciding To Take Part in a Research Study

- If you elect to participate in this study, it may delay treatment with other options such as platinum based treatment if you are platinum sensitive at this time.
- Someone will explain this research study to you.
- You can ask all the questions you want before you decide.
- Whether or not you take part is up to you.
- You can choose not to take part.
- You can agree to take part and later change your mind.
- Your decision will not be held against you.

# Why is this research being done?

Gynecological cancer that has returned (recurs) or re-grows (progresses) after surgery and/or drug therapy) rarely can be cured with standard treatments.

A healthy immune system is designed to use the body's own defenses to attack and kill foreign "invaders" such as bacteria and virus which cause infection. Cancer has a unique ability to turn off a body's normal defenses allowing cancer cells to grow and spread without detection by the immune system. As more is learned, immunotherapy (treatment that stimulates the immune system to help it fight cancer), cell therapy (introducing healthy cells into the body to replace or repair damaged cells), and targeted therapies (treatment designed to attack certain types of cells) have become new approaches in addition to surgery, radiation therapy, and chemotherapy.

This study uses two investigational agents: FT538, a cell product that stimulates the immune system into action and enoblituzumab, a monoclonal antibody (mAb) that targets an antigen found on the surface of some solid tumor cancer cells.

FT538 is a type of cell product made up of "natural killer" or NK cells. NK cells are a type of immune blood cell that are known to attack cancer cells. FT538 is produced by growing cells that come from a healthy human donor. The donor cells are treated with a process that turns them into a type of cell called an induced pluripotent stem cell, which means that these cells can be turned into any type of human cell. In this case, the cells are turned into NK cells which, once ready as FT538, are stored frozen until shipped to the study site where they are stored frozen until needed.

FT538 is different from the NK cells in your body because FT538 has been changed through a process known as cell engineering. This type of cell engineering changes the coded blueprint of cells, known as DNA, affecting how the cells work in the body. Specifically:

- A special protein called "hnCD16" has been added to FT538 so it can attach to a type of anti-cancer drug called monoclonal antibodies to help NK cells target and kill cancer cells.
- Another protein called an "IL-15/IL-15 receptor complex" has also been added to FT538.
   This helps the NK cells stay alive.
- Finally, FT538 has been engineered to remove a protein called "CD38." CD38 is naturally
  present on NK cells. Removing CD38 allows certain monoclonal antibodies that target
  CD38, to kill the cancer cells, but not to kill FT538 cells. The removal of CD38 may also
  increase the activity of NK cells.

FT538 is considered a xenotransplantation product because it comes in contact with cells of animal origin during the manufacturing process. There are risks of taking a xenotransplantation product. Refer to the sections "What are the risks of this study? Is there any way being in this study could be bad for me? (Detailed Risks)" and "What Are My Responsibilities?" for more information.

Enoblituzumab belongs to a group of drugs called monoclonal antibodies (mAB). Enoblituzumab targets cancer cells that make a lot of a protein called B7-H3. Another way to say it is that the cells "overexpress" the protein. B7-H3 is widely expressed by a number of different tumor types, including a majority of ovarian cancers. Very few normal cells express B7-H3. Enoblituzumab is thought to work by recognizing cancer cells that overexpress the B7-H3 protein and directing the body's immune system to kill those cells.

Both of these agents are considered investigational. They are not approved by the United States (US) Food and Drug Administration (FDA) for general use; however, they each were developed based on similar therapies.

Up to 6 Dose Cohorts (study groups) will be tested. The first 4 Dose Cohorts will be FT538 monotherapy (without enoblituzumab). Cohorts 5 and 6 will be FT538 plus enoblituzumab. You will be told the currently enrolling dose cohort as part of this consent discussion.

The primary purpose of this study is to identify a safe dose of FT538 cells when given alone (monotherapy) and in combination with enoblituzumab. Another purpose of this study is to gain early information on many women who have disease stabilization or shrinkage by the time of the 1st disease reassessment.

# How long will I be in this study?

Direct study participation is approximately 1 year; however, the most intensive study treatment is during the 1<sup>st</sup> 4 to 5 weeks with follow-up visits every 3 months through 1 year.

At approximately 5 weeks the computed tomography (CT) scan of the chest, abdomen and pelvis is repeated. If your disease is stable or improved from your previous CT scan, you may be offered a second course of FT538 which would require signing a separate retreatment consent form. If no further study treatment is planned and your intraperitoneal (IP) catheter is still in place, it would be removed.

<u>If you are enrolled into Dose Cohort 5 or 6</u>, enoblituzumab may continue as an intravenous infusion once every 3 weeks until it is no longer of benefit, you have unacceptable side effects, or decide to discontinue study treatment. A final study treatment visit is done approximately 4 weeks after the last dose of enoblituzumab.

<u>Follow-up visits occur every 3 months for the 1<sup>st</sup> year.</u> If you are continuing on enoblituzumab, follow-up visits will occur during a planned visit. Disease reassessments are done according to standard of care with the results documented on study case report forms.

After 1 year, you will transfer to a long-term follow-up (LTFU) study to determine if there are any late effects of FT538. FT538 is an "engineered" cell product and the FDA recommends yearly follow-up for 15 years. You will sign a separate consent form for the LTFU study. Participation in the LTFU study is required for receiving study treatment on this study.

#### What will I need to do to participate?

If you are interested in this study, you will be asked to sign this consent form giving permission to formally evaluate you for this study. This is called screening and consists of the following routine evaluations:

- Physical exam and medical history
- Routine blood work including a CA125 level (a test requiring approximately 2 teaspoons
  of blood to determine the amount of the protein cancer antigen 125)
- CT scan of your chest, abdomen and pelvis if not done in the previous few weeks
- An echocardiogram of your heart to determine cardiac function
- If you have shortness of breath or a history of lung issues, pulmonary function tests will be done

- If you had previous spread of the cancer to your brain or symptoms of possible spread, a CT or magnetic resonance imaging (MRI) of the brain will be done
- Any other tests or procedures as determined by the study doctor based on your current or past medical history

If you are eligible, a peritoneal port (a small chamber allowing access between the muscles and organs of the belly, or abdomen) and intraperitoneal catheter (a thin tube leading to the tissue of the abdomen) will be placed during an outpatient procedure in interventional radiology. It provides a painless way of withdrawing excessive fluid from the abdominal or peritoneal cavity and as a way to give the FT538 cells. The IP catheter will stay in place for at least 5 weeks.

Occasionally, because of interior scarring from previous surgeries, the catheter cannot be inserted. If it cannot be placed, you would not be eligible to continue on this study. Other treatment options would be discussed with you.

# Study Treatment is given in the following order:

- Cyclophosphamide and Fludarabine (CY/FLU) are given as IV (into a vein) infusions, one after the other, in the outpatient clinic for two days in a row.
- FT538 is given as 3 weekly doses into the IP catheter with the 1<sup>st</sup> dose no sooner than 48 hours (2 days) after the last CY/FLU dosing. Each cell infusion is given on the inpatient unit as a short stay.
- If you are enrolled in Dose Cohort 5 or 6, Enoblituzumab is given as an intravenous (into a vein IV) infusion in the outpatient clinic the day before the CY/FLU is started (although the schedule may be adjusted on an individual basis). It is given again 1 week after the last dose of FT538 and may continue every 3 weeks as long as it is of benefit.

More detailed information about the study procedures can be found under "What happens if I say yes, I want to be in this research?"

#### Is there any way that being in this study could be bad for me?

You will have side effects from the study treatment given in this study.

This study requires the placement of an intraperitoneal (IP) catheter into your abdomen to give the FT538 cells. There is risk associated with the penetration of the abdominal cavity during the IP catheter placement as it may expose new surfaces for the cancer cells to attach and grow, such as along the catheter track.

Fludarabine and cyclophosphamide are common chemotherapy drugs given in this study to prepare for the FT538 cells by blunting your immune system to lessen the chance of a reaction to the FT538 cells. The drugs will lower your blood counts (white blood cells) increasing the risk of infection.

In this study the FT538 is given into the abdomen through the IP catheter. In previous studies using similar cell products, abdominal pain and cramping was the most frequent complaint.

When FT538 is given as an IV (into a vein) infusion the most common side effects are chills and rarely, an allergic reaction. Signs of a reaction are flushing of the face, change in blood pressure and/or heart rate, difficulty breathing.

If you are in Dose Cohort 5 or 6, the most common side effect of enoblituzumab (occurring in approximately 1 out of every 2 participants) is an infusion related reaction during or shortly after the study drug is given. Signs of a reaction include fever, chills, nausea, itching, difficulty breathing and/or low blood pressure. The infusion can be slowed and/or interrupted if signs occur and medications given to reduce the severity of the reaction.

More detailed information about the risks of this study can be found under "What are the risks of being in this study? Is there any way being in this study could be bad for me? (Detailed Risks)" and in the "What happens to the information collected for the research, including my health information?" section.

# Will being in this study help me in any way?

There may be no benefit to you from participating in this research study. Your cancer may not shrink, or it may even get worse. Information learned from this study may benefit others with cancer through a better understanding of cancer and the immune system leading to future research.

What happens if I do not want to be in this research? What are my alternatives? You do not have to be in this study.

Your participation in this study is voluntary. You can decide not to be in the study and you can change your mind about being in the study at any time. There is no penalty to you, and you will not lose any benefits except for potential benefits having to do with the study.

Other options may include:

- Other investigational treatments at this institution or at another research center.
- Continue platinum based therapy, if you are platinum sensitive.
- No treatment at this time with comfort care only. This type of care helps manage pain, tiredness, appetite problems and other quality of life issues caused by the cancer. It does not treat the cancer directly, but instead tries to improve how you feel. Comfort care tries to keep you as active and comfortable as possible. If you think you might prefer comfort care, please discuss this with your family, friends and your doctor.

Your study doctor can provide you additional information, including the risks and benefits of each option.

### **Detailed Information About This Research Study**

The following is more detailed information about this study in addition to the information listed above.

## A study summary is found at the end of this document.

# How many people will be enrolled in this study?

Enrollment will most likely include 19 participants including a minimum of 10 people treated at the best tolerated Dose Cohort. Up to 33 participants may be required if side effects are seen early in the study requiring the dose cohorts to expand to 3 participants each.

# What happens if I say "Yes, I want to be in this research"?

If you are eligible and agree to take part in this study the following will occur:

**Peritoneal Port and Intraperitoneal Catheter** must be placed before any study related treatment is started.

A peritoneal port is a small reservoir or chamber that is surgically implanted under the skin to provide a painless way of withdrawing excess fluid or delivering anti-cancer drugs into the abdominal or peritoneal cavity over a period of weeks or longer. The port has a silicone rubber top that can be penetrated by a needle and an attached catheter that is designed to hang down into the abdominal cavity once it is placed inside the body. The port is placed underneath the skin and then sutured (stitched) to the ribs.

The port and IP catheter are placed during an outpatient procedure in Interventional Radiology. Numbing medication and other medications will be used to reduce the pain. You will experience pain at the site of insertion until it heals.

Occasionally, because of adhesions (internal scarring of tissue or organs) from previous surgeries, the catheter cannot be inserted. If it cannot be placed, you would not be eligible to continue on this study. Other treatment options would be discussed with you.

**Cyclophosphamide and Fludarabine (CY/FLU)** are given as IV infusions, one after the other, in the outpatient clinic for two days in a row. Each infusion takes about 30 minutes, although fluids and medications are given before and after the infusion, so it will take longer than the 1 hour study drug infusion time.

**FT538** is given as 3 weekly doses into the IP catheter with the 1<sup>st</sup> dose no sooner than 48 hours (2 days) after the last CY/FLU dosing. Each study treatment is given on the inpatient unit as a short stay. The FT538 is infused quickly (by gravity) followed by flushing of the tube with fluids. Depending on your dose, it may be given as one or more bags of cells. After the FT538 infusion, you will be asked to change positions every 15 minutes for 2 hours to distribute the cells throughout your abdomen.

Three days after the 1st FT538 infusion only, you will have a clinic appointment with bloodwork.

FT538 is given weekly in a manner identical to the first infusion, on Day 1, Day 8 and Day 15.

## If you are assigned to Dose Cohort 5 or 6 (FT538 plus enoblituzumab):

The first dose of enoblituzumab is given as an intravenous (into a vein – IV) infusion over approximately 2 hours in the outpatient clinic.

A second dose is given approximately 1 week after your last FT538 infusion.

As described in the next section, a repeat CT scan of the chest, abdomen and pelvis is done around this same time. If the CT scan shows stable or shrinking disease, enoblituzumab may continue once every 3 weeks as an outpatient IV infusion for up to 1 year unless unacceptable side effects occur or your disease worsens.

Routine bloodwork and a clinic visit will occur with each study treatment. A final study treatment visit will be done approximately 4 weeks after your last dose of enoblituzumab for a routine exam and blood work to ensure there are no ongoing side effects.

# Visits and repeat CT scan after the 3rd FT538 infusion:

After the last FT538 infusion you will return to clinic once a week for 4 weeks for a clinic visit, assessment of side effects, and routine blood work. If enoblituzumab is scheduled, the appointments will be scheduled on the same day if possible.

Approximately 5 weeks after the 1st dose of FT538 infusion a repeat CT scan of the chest, abdomen and pelvis will be done. If it shows stable or shrinking disease, you may be offered a 2nd study treatment course (identical to the 1st). If you plan on a 2nd course, your IP catheter will remain in place. If a second course of FT538 is not planned, your IP catheter will be removed as soon as the decision is made.

## Disease Re-Assessment and study visits through 1 year

You will continue with routine follow-up imaging studies and CA-125 levels every 3 months. A follow-up visit is required at 3, 6, 9 and 12 months after the 1st FT538 infusion. If you are continuing on enoblituzumab, the follow-up visit will be aligned with one of those visits.

# Long-term follow-up after 1 year

FT538 is a genetically engineered cell product and the FDA is recommending follow-up for up to 15 years from the 1st dose. This follow-up can be done in person if you are receiving care at the University of Minnesota. Otherwise it can be done by phone, email or mail. You will be required to sign a separate consent for the long-term follow-up (LTFU) study.

# STUDY RELATED SAMPLE COLLECTION (RESEARCH RELATED):

As this is a clinical research study, additional blood is collected for research related testing (70 ml or about 5 tablespoons) at key time points and up to 3 additional time points if felt important on an individual basis to learn about individual differences (for example, in the case of a very good disease response, unexpected side effects):

- Before study treatment starts
- Before the 1<sup>st</sup> dose of enoblituzumab if you are enrolled in Cohort 5 or 6

- Before the 1<sup>st</sup> CY/FLU study treatment
- Before each FT538 infusion
- At the clinic appointment approximately 3 days after the 1<sup>st</sup> dose of FT538
- At each weekly visit after the FT538 infusion
- At the 3, 6, 9, and 12 month follow-up visits (approximately 40 milliliters or about 3 tablespoons) if you have a worsening of your disease or start a new treatment, these samples may not be collected.

Approximately 2 teaspoons of blood of additional blood will be collected around the time of your disease reassessment for to look for evidence of an immune response to FT538.

In addition, approximately 2 teaspoons of blood is collected at the 3, 6, and 12 month follow-ups and sent to Fate Therapeutics as part of their long-term follow-up testing required by the FDA. These samples are stored frozen and shipped in batches to Fate Therapeutics for testing required on their products by the FDA.

Participation in this study involves collection of blood that may result in a decrease in your overall hemoglobin level and may require a whole blood transfusion. Please speak to your study doctor if you have questions.

The research blood samples will be analyzed to look at changes in your immune system over time, the effects of the study drugs (FT538, and if receiving, enoblituzumab), and how long the study drugs are present in your blood. Testing may include analysis of your genome (DNA), which is the "instruction book" for the cells in your body. Your samples may be tested to find out about mutations (permanent changes) and other possible changes to your genome. Testing will not be done to determine whether any of the mutations are inherited.

Fluid will be collected from your abdomen through your IP catheter for research related analysis. Samples will be collected at the time your IP catheter is placed, prior to each FT538 infusion, and once a week until FT538 cells are no longer detected (approximately 2 weeks after the last FT538 infusion) and at the catheter removal. If you have ascites (fluid pooling in your intraperitoneal space as a result of the cancer), these cells will be used. Otherwise, cells are obtained by an intraperitoneal (IP) washing where a small amount of normal saline is infused through your IP catheter. You then are asked to move around to distribute the fluid and then it is withdrawn through your IP catheter. Approximately ¼ cup of fluid is needed, but if more is available (as in the case of ascites), more will be collected.

If feasible, a sample of tumor tissue will be taken by biopsy when your IP catheter is placed and at the time the IP catheter is removed. Your safety comes first - the biopsies are done only if tumor is easily accessible.

At the time of study enrollment you are assigned a unique participant code that will be used instead of your name or other identifying information. The research samples are labelled with your unique code making it difficult for anyone looking at the sample to know it belongs to you.

Research related testing is primarily done at the University of Minnesota and M Health /Fairview laboratories; however, for specialized testing that cannot be done within the system, samples may be sent to outside laboratories, including Fate Therapeutics, and if receiving enoblituzumab, MacroGenics. Any samples sent outside of the system is labelled with the unique participant code assigned at enrollment.

None of the research related testing results will affect your care or your participation in this study. Neither you nor your health insurance provider will be charged for the cost of research sample collection, processing, storage, and testing.

There may be some leftover cells from the samples collected for research purposes. With your permission, after analysis for this study is completed we would like to store any leftover samples for future analysis as new research tests become available. They will not be used for studies other than ones to learn about the immune system and/or cancer. You will be asked to indicate your decision about future use of leftover samples at the end of this document.

## **New findings**

Any new important information that is discovered during the study which may influence your willingness to continue participation in the study will be provided to you.

## What are my responsibilities?

Because FT538 is a xenotransplantation product, you are also expected to have certain responsibilities in the future. These future responsibilities may include, but are not limited to, having regular check-ups and telling your doctor or other healthcare providers about receiving a xenotransplantation product in the event of unexplained illnesses. You and your family members and intimate contacts should not donate blood, sperm, or other body fluids or tissues. If needed, ask the study doctor or a member of the study staff to help you discuss this with your family members and intimate contacts, or if you have any questions.

## What happens if I say "Yes" but I change my mind later?

If you take part in this research study, and want to leave, you should let a member of the research team or your study doctor know. Your choice not to be in this study will not affect your right to any present or future medical care.

If you leave the study before the planned final visit, you may be asked by the study doctor to have some tests or procedures for your safety.

The study doctor may stop your participation in this study at any time without your consent for reasons including the following:

- It appears being in the study may be harmful to you;
- There is a change in the research and/or the risk profile that requires your re-consent and you refuse to sign the updated consent form;
- If the study is stopped early.

If you end participation in this study early, the information about you, test results, and laboratory samples that were collected while you were participating in the study may still be used. Follow-up information will still be requested unless you withdraw consent.

# What are the risks of being in this study? Is there any way being in this study could be bad for me? (Detailed Risks)

## Risks of being in this study:

You will experience side effects. You may experience all, some, or none of these side effects and the side effects may vary in severity. The severity may be mild, moderate, or severe, up to and including death. Also, there is always the risk of a rare or previously unknown side effect occurring.

This multi-day study therapy may trigger or worsen underlying conditions such as a fast and irregular heartbeat (atrial fibrillation/flutter), chronic obstructive pulmonary disease (COPD), or may make management of chronic conditions such as hypertension (high blood pressure) or diabetes more difficult during study therapy.

The University Of Minnesota has been doing studies with NK cells similar to this study for several years including by intraperitoneal administration; however this is an early study of FT538 in humans and the 1<sup>st</sup> as an intraperitoneal infusion, so its side effects are not well documented.

Other drugs will be given to make side effects less serious and uncomfortable or your study doctor may delay or alter the planned study treatment. Many side effects go away shortly after the study drugs are stopped, but in some cases side effects can be serious, long-lasting or permanent, even fatal.

Cyclophosphamide (CY) and fludarabine (FLU) are commonly used chemotherapy drugs and are available without being on a research study.

# Risks Related to Cyclophosphamide (CY)

CY may cause side effects, as described below.

| Common Side Effects - occurring in more than 30 out 100 participants receiving this drug | |
|---|---|
| <ul> <li>Low blood counts: Your white and red</li> </ul> | Nausea and vomiting (more common with |
| blood cells and platelets may temporarily | larger doses) |
| decrease. This can put you at increased risk | Temporary hair loss |
| for infection, anemia, and/or bleeding. | Discoloration of the skin or nails |
| Poor appetite | |
| Less Common Side Effects - occurring in about 10 to 29 participants receiving this drug | |
| Loss of fertility | Bladder problems and bleeding |
| Diarrhea | (hemorrhagic cystitis) |
| Mouth sores | |

Serious, but uncommon, side effects of CY include:

- Increased risk of developing other cancers, such as bladder cancer, acute leukemia (a type of blood cancer), lymphoma (a type of lymph node cancer), thyroid cancer, and/or sarcoma (a type of cancer that can start in the soft tissue, bone, or other tissue).
- Liver problems, which can be fatal
- Heart failure, which can be fatal
- Inflammation of the lung

CY may cause rare and unexpected side effects other than those described here. Tell the study doctor if you have any unusual problems while receiving this study drug.

## Risks Related to Fludarabine (FLU)

FLU may cause side effects, as described below.

| Common Side Effects (occurring in more than 30% of participants) | |
|---|---|
| Fever | Poor appetite |
| Infection | Low blood counts. Your white and red |
| Weakness | blood cells and platelets may temporarily |
| Cough | decrease. This can put you at increased risk |
| Nausea and vomiting | for infection, anemia, and/or bleeding. |
| Less Common Side Effects (occurring in about 10%-29% of participants) | |
| • Chills | <ul> <li>Shortness of breath (lung problems)</li> </ul> |
| Fatigue | Diarrhea |
| • Pain | Rash (skin reactions) |
| Sweating | Swelling |
| <ul> <li>Numbness and tingling of hands and feet</li> </ul> | Taste changes, metallic taste |

# Serious, but uncommon, side effects of FLU include:

- An increased risk of infection (such as herpes, fungal infection, and a type of pneumonia that occurs in people with weakened immune systems called *Pneumocystis carinii*) due to suppression of the immune system
- Severe side effects involving the brain and other parts of the nervous system, which were seen at doses higher than the dose you will receive in this study
- Hemolytic anemia (destruction of red blood cells)
- A rare condition called transfusion-associated graft-versus-host disease (also called GvHD), which occurs when immune cells in a blood transfusion attack cells in the body causing fever, rash, liver problems, and abdominal pain and diarrhea. If you require a blood transfusion while on this study, you will receive only blood transfusions that have received radiation treatment to reduce the risk of transfusion-associated GvHD.
- Tumor lysis syndrome (also called TLS) can happen when cancer cells have broken down
  and byproducts of that breakdown have entered the bloodstream. Symptoms may
  include weakness, low blood pressure, muscle cramps, and decreased urination. TLS can
  lead to kidney damage and/or other organ damage. In addition to cancer treatment,
  many factors including the type and extent of the cancer, as well as treatments given to

an individual, can contribute to TLS. Let the study doctor know immediately if you develop these symptoms.

FLU may cause rare and unexpected side effects other than those described here. Tell the study doctor if you have any unusual problems while receiving this study drug.

# Risks of FT538

FT538 has not been widely used in humans and has only been given as an intravenous (IV - into a vein) infusion.

In this study, the FT538 is given directly into the abdominal space through an IP catheter. This is the first time that FT538 is being given as an intraperitoneal infusion, and therefore the risks are not known. In previous studies using similar cell products given intraperitoneally (IP), abdominal cramping was the most frequent complaint. You will be given acetaminophen (Tylenol®) and diphenhydramine (Benadryl®) before the FT538 infusion and every 4 hours afterwards as needed. In some situations abdominal pain and cramping has required stronger oral or intravenous pain control.

Risks of FT538 based on intravenous (IV) infusion are listed below:

The potential risks of FT538 based on IV infusion include those related to how FT538 may work in the body and how the body may react to FT538. The potential side effects listed below are based on laboratory studies and knowledge of similar cell therapies.

- An infusion related (allergic) reaction during or shortly after the FT538 cell infusion.
  There is a potential risk for an allergic reaction during intravenous (IV) infusion. The
  reaction with IV infusion may be mild (skin irritation/rash) to life-threatening (difficulty
  breathing/swelling of the face and throat). Please seek treatment immediately and tell
  the study doctor and research team if you have any of these symptoms, or any other
  side effects, during the study.
- Cytokine release syndrome (CRS) is a serious systemic (whole body) inflammation
  response. CRS is seen with other types of cell therapies, but is not typically seen with NK
  cell therapies. Signs of CRS include fever, nausea, headache, rash, rapid heartbeat, low
  blood pressure, and trouble breathing. Most patients who develop CRS have a mild
  reaction, but sometimes, the reaction may be severe or life threatening. CRS is treated
  with supportive care and steroids.
- Tumor lysis syndrome (also called TLS) can happen when cancer cells have broken
  down and byproducts of that breakdown enter the bloodstream. Symptoms may include
  weakness, low blood pressure, muscle cramps, and decreased urination. TLS can lead to
  kidney damage and/or organ damage. In addition to cancer treatment, many factors can
  contribute to TLS, including the type and extent of a patient's cancer, as well as
  treatments given to a patient. Let your study doctor know immediately if you are unable
  to urinate.
- Effect on the nervous system have been seen with other types of cell products, but is not a common risk of NK cell therapies. Neurotoxicity (when substances alter normal

- activity of the nervous system) symptoms observed with other cell therapies include confusion, delirium, and sometimes seizures and cerebral edema (swelling) that could lead to death. You will be monitored for changes in your mental status before and at every clinic visit after FT538.
- **Reaction to DMSO** (dimethyl sulfoxide) is a common ingredient in cell therapy products. Some people have a negative reaction to DMSO. If you have had a previous reaction related to DMSO, you will not be eligible to take part in this study. Because of the very small volume of the cell infusion and it is given into your abdominal space, no reaction is expected. DMSO may cause side effects like coughing, flushing, rash, chest tightness, wheezing, nausea, vomiting, and high or low blood pressure.
- There is an increased risk of infection. FT538 contains cells from human donors and
  may transmit infectious diseases or infectious agents, such as viruses, bacteria, or other
  pathogens, and/or other non-infectious agents, which may also cause side effects. The
  master cell bank from which FT538 is manufactured has been extensively tested to
  reduce the risk of disease infection. However, these tests do not completely eliminate
  this risk. For some infectious agents, there are no routine tests to predict or prevent
  their presence.

There may be other risks that are unknown which could range from mild to serious, and even fatal. The use of NK cell products like FT538 is investigational.

## **Risks Related to Xenotransplantation Products**

FT538 is considered a xenotransplantation product because it comes in contact with cells of animal origin (mouse cell) during the manufacturing process. Risks of receiving a xenotransplantation product may include, but are not limited to, developing infections from agents that may be associated with cells of animal origin, transmitting these infectious agents to others, and the growth of tumors. The animal cells, which come into contact with the FT538 cells during the manufacturing process, originate from a master cell bank that has been extensively tested to reduce these risks. However, these tests do not completely eliminate this risk. The likelihood and timing for developing a condition or illness from xenotransplantation products is unknown. If you have any questions about the risks involved in receiving a xenotransplantation product, ask the study doctor or a member of the study staff.

**FT538** has been genetically engineered (the structure of the NK cell has been changed from the state in which NK cells naturally exist in your body) using virus-based technology. The long-term risks of the genetic engineering and the viruses used to make these changes are not known. As a result, the FDA requires long-term follow-up at least once a year for up to 15 years. Of interest is the development of cancer, new or worsening neurologic disorders, new or worsening autoimmune (immune reactions) or rheumatologic (of the immune system) disorder, or new blood disorder. Details of the long-term follow-up study are provided in a separate consent form.

# Risks of Enoblituzumab (Dose Cohorts 5 and 6 only) General risks associated with drugs similar to enoblituzumab:

- Infusion reactions: These are generally temporary reactions. They usually happen during or within hours after getting the study drug. A mild to moderate reaction can cause a fever, chills, nausea, vomiting, headache, confusion, seizures, muscle stiffness, rash, or itching. A more severe infusion reaction can also cause low blood pressure, and difficulty breathing. They can be life threatening, cause hospitalization, or rarely may cause death.
- Immune-related side effect: A possible side effect of the test drug is that your immune system may attack other, healthy parts of your body. This is known as an autoimmune reaction. This reaction can affect many different organs in your body. If you have a reaction, you may require treatment with high-dose steroids or hospitalization. Patients who have received other drugs that affect the immune system have experienced the following types of side effects:
  - Pneumonitis (inflammation in the lungs): Symptoms may include shortness of breath, chest pain, and/or cough.
  - Colitis (inflammation of the colon): This may lead to tears or holes in your colon (large intestine). Symptoms may include diarrhea or more frequent bowel movements, black or tarry stools (that may have blood or mucous), and/or severe abdominal pain.
  - Hepatitis (inflammation of the liver): Symptoms include yellowing of your skin or the whites of your eyes. You might have nausea or vomiting, abdominal pain, and feel less hungry than usual. Other signs include fevers or chills, dark urine, and/or bleeding or bruising more easily than usual.
  - O Hormone gland problems (including thyroid, pituitary [pituitary gland is a gland in the brain that produces hormones], adrenal and pancreas): If you have hormone gland problems, you might feel a rapid heartbeat, have changes in weight, or increased sweating. You may feel hungrier or thirstier than usual. You may need to use the toilet more often. Other possible side effects are hair loss, feeling cold, constipation, deeper voice, muscle aches, dizziness or fainting, and/or unusual headaches.
  - Kidney problems: Symptoms may include changes in the amount or color of your urine, swelling of ankles, and/or loss of appetite.
  - o **Encephalitis (inflammation of the brain):** You may feel headache, fever, tiredness, and confusion. You might have memory problems, weakness, see or hear things that are not there, uncontrolled muscle movements, and/or stiffneck.
  - Skin problems, including Stevens-Johnson syndrome (SJS) and toxic epidermal necrolysis (TEN): Inflammation of the skin so you may have widespread peeling of the skin, itching, and redness. More severe inflammation of the skin may involve the inside of your mouth, the surface of your eye, genital areas, and/or may cause the top layer of your skin to peel from all over your body, which may cause severe, potentially life-threatening, infection.
  - Myocarditis (inflammation of the heart muscle): Inflammation of the heart muscle may cause difficulty pumping your blood throughout your body. This can result in

- chest pain, shortness of breath, swelling of the legs, fast or irregular heartbeat and/or dizziness or fainting.
- o **Problems in other organs:** You might have changes in eyesight, severe muscle or joint pain or weakness, and/or low red blood cells (anemia).

#### Enoblituzumab

As of April 2021, 349 adult participants had received enoblituzumab at doses up to 15.0 mg/kg, which is the dose given in this study.

So far, the most important safety risk that has been identified with enoblituzumab is infusion-related reaction (IRR), including reactions known as cytokine release syndrome (CRS). IRRs are effects due to a drug that may occur during or shortly after an infusion. Signs and symptoms of an infusion-related reaction may include:

- fever
- chills
- nausea
- vomiting
- headache
- muscle stiffness
- rash
- itching
- low blood pressure
- difficulty breathing

IRRs can be life threatening and, in rare cases, may cause death. For all adult studies, IRRs (including CRS) have occurred in 48% of participants receiving study treatment with enoblituzumab. Most of the infusion-related reactions observed in participants receiving enoblituzumab have been mild to moderate in severity with 6 % of participants having more severe infusion-related reactions (including two who experienced life-threatening IRR events). These participants, some of whom were hospitalized for these reactions, recovered after receiving treatment with steroids, antihistamines and intravenous fluids.

The following were the most common side effects that were considered related to enoblituzumab administration and were seen in at least 1 of 10 adult participants. These side effects have been generally mild or moderate.

- infusion related reactions (described above)
- fatigue
- nausea
- chills
- vomiting

Eleven (11) participants have experienced serious side effects that were considered related to enoblituzumab. Serious side effects that occurred in 3 or more participants included:

IRRs

## Risks of the Peritoneal Port and Intraperitoneal (IP) Catheter Placement and Use

Rarely, a complication can occur at the time of IP catheter placement due to the bowel being stuck to the abdominal wall from scar tissue formed during prior surgery. The risks of placement of the IP catheter include infection, bleeding and damage to surrounding organs such as the bowel. If the interventional radiologist does not feel that they can safely place the catheter, the procedure will be terminated and you will not be able to receive study treatment under this study. Sometimes these IP catheters are placed and they do not function well, but this is uncommon.

There is a risk that cancer cells that are located within the peritoneum could spread to surrounding tissues such as the abdominal wall. This risk is associated with the penetration of the abdominal cavity during the IP catheter placement as it exposes new surfaces for the cancer cells to attach. Implantation of cancerous cells within surgical incisions, along biopsy needles and drainage catheter tracts is a recognized mechanism for the spread of cancer. Instances of this happening have been reported in the literature. Spread of cancer cells is a potential hazard of all invasive procedures in the case of any malignancy. Although this is thought to be a rare event, placement of an IP catheter in your abdomen may put you at risk for tumor cells spreading to surrounding tissues.

The plan is to keep the IP catheter in place until around Day 36 (after the repeat CT scan of the chest, abdomen, and pelvis) or once it is determined that you will not be retreated. The primary risk associated with keeping an IP catheter in for any period of time is localized skin infection. Although this risk is rare (less than 1%) it would require antibiotic treatment. Very rarely, the catheter becomes plugged. The catheter would be removed early if it posed a risk or was not functional.

#### **General Risks of Intraperitoneal Infusions and Washings**

- abdominal discomfort due to the infusion of fluids into the abdominal area
- fever
- infection within the abdomen

### **Risks of Intraperitoneal Biopsy**

The biopsies will be done in Interventional Radiology (where the IP catheter is placed) and will only be done if tumor cells are easily accessible. Risks may include:

- You will have an injection of a local anesthetic to numb the area where the biopsy will be taken it stings for a moment before the area goes numb. After that you only feel mild to moderate pressure as the biopsy is taken.
- Slight risk of bleeding which usually requires no treatment overall of all types of ultrasound/CT guided biopsies 1-2 participants out of 1,000 experience bleeding.
- Slight risk of infection

The biopsy site may be uncomfortable for a day or two

#### **Risks of Routine Tests and Procedures**

#### Risks of Blood Collection

Risks of having blood drawn for routine blood tests and research purposes include:

- pain at the site of the needle stick
- tenderness and/or bruising at the site of blood collection
- dizziness, light-headedness, rarely fainting
- very rarely, infection at the site of the needle stick

## Risks of a chest, abdomen, pelvis CT scan or Positron Emission Tomography (PET)/CT

A CT scan is a computerized x-ray picture of your internal organs. You may feel some discomfort or anxiety when lying inside of the CT scanner.

A PET scan helps doctors see changes due to certain disease in organs and tissues inside your body. A PET scan may cause you to feel "closed in" while lying in the scanner. However, the scanner is open at both ends and an intercom allows you to talk with doctors and staff. If you feel ill or anxious during scanning, doctors and/or technicians will give comfort or the scanning will be stopped. The PET scan exposes your body to radiation. The radioactive solution does not remain in your system for a long period of time. However, you should wait 2 hours before holding an infant or getting close to a pregnant woman to avoid exposing them to radiation. You should drink fluids after the scan to help remove the solution from your system.

You will be exposed to ionizing radiation during the scanning to evaluate your disease status. The scientific unit of measurement for radiation dose is the millisievert (mSv). The average amount of radiation received from natural sources of radiation by a Minnesota resident in one year is 3 mSv. Each CT scan of the chest, abdomen and pelvis would expose you to 18 mSv radiation. This is equal to approximately 5.6 years of background radiation. If you have a PET/CT each exposure is 25 mSv and equal to approximately 8.3 years of background radiation. Exposure to radiation may increase your lifetime risk of developing a 2<sup>nd</sup> cancer. If you have additional questions, you may ask your study doctor.

Your disease re-assessment study may be done with CT contrast (a chemical substance to allow a better view of what is being scanned). Your study doctor can tell you if the dye is necessary for your procedure. The contrast material (dye) that is injected into your body may cause you to get a metallic taste in your mouth and to feel warm. Rarely, it causes nausea and vomiting. You may develop a skin rash or itchiness if you're allergic to the contrast. A life-threatening allergic reaction can also happen, but this is rare. Tell your study doctor about any sensitivities to medications, or any kidney problems you have. IV contrast can increase the risk of kidney failure if you're dehydrated or have a pre-existing kidney problem.

#### Risks of MRI

During the MRI, you may feel mild vibrations throughout your body. The machine will produce a loud knocking noise. This is normal. You will be given earplugs to protect your ears. Some

people, especially those who tend to feel uncomfortable in small or closed spaces, may feel "closed in" and become anxious while in the scanner. The scanner has an intercom, which will allow you to speak to the staff during the procedure. If you feel ill or anxious during scanning, tell the MRI staff and the scanning will be stopped if you wish. The magnetic field used in MRI scanning may harm people who have metal in their bodies (pacemakers, neurostimulators, certain clips, or staples from surgery). It may cause problems with devices, such as pacemakers. If you have metal in your body or a pacemaker, you should not have an MRI.

## Risks of Echocardiogram (ECHO)

There are no known risks from an echocardiogram (ECHO) because the test uses only sound waves to evaluate your heart. These high-frequency sound waves have not been shown to have any harmful effects.

## Risks of Ultrasound used for the IP catheter placement and removal

There is little risk associated with ultrasound – there is no ionizing radiation exposure associated with ultrasound imaging. Ultrasound waves can heat the tissues slightly. In rare cases, it can also produce small pockets of gas in body fluids or tissues (cavitation).

### Risks of Pulmonary Function tests

You may have some coughing or experience some shortness of breath after the pulmonary function test, but there is no pain associated directly with these tests.

#### Other Risks:

- Risks of Genetic Research The risks to you and your family from genetic research on the blood samples are very low. The unique participant code assigned at study enrollment is used instead of your name or other identifying information making it difficult for anyone looking at the sample to know it belongs to you. Testing is done in batches (more than 1 participant at a time) and no research results will be placed in your medical record.
- Because this study involves the use of your identifiable, personal information, there is a
  chance that a loss of confidentiality will occur. There are procedures in place to lessen
  the possibility of this happening (see "What happens to the information collected for
  the research, including my health information?" section below).

# Reproductive Risks: If you are able to become pregnant (pre-menopausal and have a uterus and ovaries) the following applies to you:

- You must have a negative pregnancy test within 14 days of the study treatment start as pregnant women cannot take part in this study.
- You must agree to use a highly effective form of contraception for at least 12 months after the last dose of cyclophosphamide or at least 4 months after the last dose of FT538.
  - If you receive enoblituzumab and continue it for more than 12 months after the last dose of cyclophosphamide, effective contraception must be used for the duration of enoblituzumab study treatment.

According to the World Health Organization and the United States Center for Disease Control and Prevention, the most effective forms of birth control include complete abstinence, surgical sterilization (both male and female), intrauterine devices (IUDs), and the contraceptive implant. The next most effective forms of birth control include injectables, oral contraceptive pills, the contraceptive ring, or the contraceptive patch. Acceptable, but least effective, methods of birth control include male condoms (with or without spermicide) and female condoms.

# Will it cost me anything to participate in this research study?

FT538 is provided at no cost by Fate Therapeutics for the purpose of this study. If you are assigned to enoblituzumab, MacroGenics will provide this study drug without cost. The cost of processing and testing any samples collected for research is paid for by study funds.

You and/or your insurance company will be billed for any standard medical care given during this research study. This means your insurance company will be billed for the placement and removal of the intraperitoneal catheter, the cyclophosphamide and fludarabine, outpatient clinic visits, the hospitalizations, routine medical care, all laboratory tests done for standard safety assessment, and assessments that are done for your medical care. You will be responsible for any copays your insurance normally issues for these visits/procedures.

# **Compensation for Participation**

You will not receive any monetary compensation for your participation in this study.

# What happens to the information collected for the research, including my health information?

The researchers will do their best to make sure that your private information is kept confidential. Information about you will be handled as confidentially as possible but participating in research may involve a loss of privacy and has a potential for breach of confidentiality. Study data will be physically and electronically secured. As with any use of electronic means to store data, there is a risk of breach of data security.

### Overview

If you participate in this study, your information, including your health information, will be used and shared for purposes of conducting this research. As described later in this Consent Form, your information may also be used and shared for publishing and presenting the research results, future research. If you sign and date this Consent Form, you are giving permission to use and share your health information for these purposes and you are giving permission to any health care providers who are treating you to share your medical records with us.

## What health information will be made available?

Health information about you to be used and shared for the research includes those items checked by the research team below:

- ☑ Your medical records, which may include records from hospital and clinic visits, emergency room visits, immunizations, medical history and physical exams, medications, images and imaging reports, progress notes, psychological tests, electroencephalography (EEG), electrocardiogram (ECG), and echocardiogram (ECHO) reports, laboratory and pathology reports, dental records and/or financial records. These records may be used and shared for as long as this research continues.
- ☑ Information collected as part of this research study, including research procedures, research visits, and any optional elements of the research you agree to, all as described in this Consent Form. This information might not be part of your medical record, and may include things like responses to surveys and questionnaires, and information collected during research visits described in this Consent Form.

## What about more sensitive health information?

Some health information is so sensitive that it requires your specific permission. If this research study requires any of this sensitive information, the boxes below will be marked and you will be asked to initial to permit this information to be made available to the research team to use and share as described in this Consent Form.

| ☐ My drug & alcohol abuse, diagnosis & treatment records (initial | I) |
|-------------------------------------------------------------------|----|
| ☑ My HIV/AIDS testing records (initial) | |
| ☐ My genetic testing records (initial) | |
| ☐ My mental health diagnosis/treatment records (initial) | |
| ☐ My sickle cell anemia records (initial) | |

#### Who will access and use my health information?

If you agree to participate in this study, your information will be shared with:

- The University of Minnesota research team and any institutions or individuals collaborating on the research with us;
- The study doctor and study staff may share your information with representatives of the University of Minnesota and M Health. These people may use your information to provide oversight and administrative support for the research, conduct evaluations and reviews, and perform other activities related to the conduct of the research;
- The University of Minnesota and representatives of this institution and its affiliates, including those that have responsibilities for monitoring or ensuring compliance, such as the Quality Assurance Program of the Human Research Protection Program.
- The research sponsor(s), any affiliates, partners or agents of the sponsor(s) involved in the research, organizations funding the research, and any affiliates, partners or agents of the funding organization(s) involved in the research;
- Organizations who provide accreditation and oversight for research and the research team, and others authorized by law to review the quality and safety of the research

(such as U.S. government agencies like the Food and Drug Administration, the Office of Human Research Protections, the Office of Research Integrity, or government agencies in other countries); and

 Advarra IRB, the independent external Institutional Review Board that is responsible for the review of this study.

Fate Therapeutics (and MacroGenics if you receive enoblituzumab) will be provided copies of any serious adverse event reports as they occur with direct identifiers removed.

## How will my information be used in publications and presentations?

Your health data will be used to conduct and oversee the research. We may publish the results of this research in scientific, medical, academic or other journals or reports, or present the results at conferences. Information that makes it easy to identify you (such as your name and contact information, social security number (SSN) and medical records number) will not be part of any publication or presentation. If you have an extremely unique or rare condition that is not shared by many others, it is possible that some people may be able to determine your identity even without these identifiers.

## Optional Consent for Future Use of Identifiable Data or Specimens

At the completion of this research study, we would like to store and be able to use and share your identifiable research related samples and/or health information with researchers at the University or affiliated hospitals for other research. Any research that involves identifiable information will be reviewed by an Institutional Review Board (IRB), which is the committee that provides ethical and regulatory oversight of research at the University, prior to use. Because these specimens and/or health information are identifiable, we are asking your permission to store, use and share these for other research.

We may not ask for your consent before using or sharing your identifiable specimens or data. You will not receive any results or financial benefit from the future research done on your specimens or data. We may share your identifiable specimens or data with outside researchers who will use them for future research. Samples are labelled with your unique study code assigned at study enrollment and information such as the date of collection/study day that can be linked back to your health information through a master study list.

If you leave the study, you can ask to have the data collected about you removed or the samples destroyed. You can also ask us to remove information that identifies you from the data or samples. This may not be possible if your samples and data have already been shared.

# Do I have to sign and date this Authorization and give my permission to make my information, including my health information, available for use and sharing?

No, you do not have to sign and date this Authorization. But if you do not sign and date it, you will not be able to participate in this research study. Treatment available outside of the study, payment for such treatment, enrollment in health insurance plans and eligibility for benefits will not be impacted by your decision about signing and dating this Authorization.

# Does my permission for making my health information available for use and sharing ever expire?

No, there is no expiration date.

May I cancel my permission for making my health information available for use and sharing? Yes. You may cancel your permission at any time by writing to the study doctor at the address on the first page of this Form. If you cancel your permission, you will no longer be in the research study. You may also want to ask someone on the research team if canceling will affect any research-related study treatment. If you cancel your permission, any health information about you that was already used and shared may continue to be used and shared for the research study and any optional elements of the study to which you agree in this Authorization.

### What happens to my health information after it is shared with others?

When we share your information with others as described in this Authorization, privacy laws may no longer protect your information and there may be further sharing of your information.

## Will I be able to look at my records?

It is possible that the research team may not allow you to see the information collected for this study. However, you may access any information placed in your medical records after the study is complete.

# What will be done with my data and specimens when this study is over?

We will use and may share data and/or specimens for future research. They may be shared with researchers/institutions outside of University of Minnesota. This could include for profit companies. We will not ask for your consent before using or sharing them. We will remove identifiers from your data and/or specimens, which means that nobody who works with them for future research will know who you are. Therefore, you will not receive any results or financial benefit from future research done on your specimens or data. No results from research related testing will be placed in your medical record.

Research samples may be sent to an outside laboratory for testing (including to Fate Therapeutics and MacroGenics, if you are assigned to enoblituzumab) that cannot be routinely performed at the University of Minnesota and M Health/Fairview laboratories. No information to directly identify you will be provided on these samples.

#### Will I receive research test results?

No, individual tests results will not be shared with participants. Research related testing is not done in real-time like laboratory work for medical care. Instead the samples are stored frozen and tested in batches at a future date.

## Whom to contact about this study:

During the study, if you experience any medical problems, suffer a research-related injury, or have questions, concerns or complaints about the study such as:

Whom to contact in the case of a research-related injury or illness;

- Payment or compensation for being in the study, if any;
- Your responsibilities as a research participant;
- Eligibility to participate in the study;
- The study doctor's or study site's decision to withdraw you from participation;
- Results of tests and/or procedures;

# <u>Please contact the study doctor at the telephone number listed on the first page of this consent document.</u>

If you seek emergency care, or hospitalization is required, alert the treating physician that you are participating in this research study.

An institutional review board (IRB) is an independent committee established to help protect the rights of research participants. If you have any questions about your rights as a research participant, and/or concerns or complaints regarding this research study, contact:

By <u>mail</u>:

Study Subject Adviser Advarra IRB 6100 Merriweather Drive, Suite 600 Columbia, MD 21044

• or call **toll free**: 877-992-4724

• or by <u>email</u>: <u>adviser@advarra.com</u>

Please reference the following number when contacting the Study Subject Adviser: <u>Pro00065732</u>.

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You may search this Web site at any time.

This research has also been reviewed and approved by an IRB within the Human Research Protections Program (HRPP) at the University of Minnesota. To share feedback privately with the University of Minnesota HRPP about your research experience, call the Research Participants' Advocate Line at 612-625-1650 (Toll Free: 1-888-224-8636) or go to z.umn.edu/participants. You are encouraged to contact the HRPP if:

- Your questions, concerns, or complaints are not being answered by the research team.
- You cannot reach the research team.
- You want to talk to someone besides the research team.
- You have questions about your rights as a research participant.
- You want to get information or provide input about this research.

## Will I have a chance to provide feedback after the study is over?

The University of Minnesota HRPP may ask you to complete a survey that asks about your experience as a research participant. You do not have to complete the survey if you do not

want to. If you do choose to complete the survey, your responses will be anonymous. If you are not asked to complete a survey, but you would like to share feedback, please contact the study team or the University of Minnesota HRPP.

# What happens if I am injured while participating in this research?

In the event that this research activity results in an injury, treatment will be available, including first aid, emergency treatment and follow-up care as needed. Care for such injuries will be billed in the ordinary manner to you or your insurance company. If you think that you have suffered a research-related injury, let the study doctor know right away. By signing and dating this document, you will not lose any of your legal rights or release anyone involved in the research from responsibility for mistakes.

## **Optional Storing of Leftover Samples for Future Research:**

Once the research associated with this study there may be some leftover blood, ascites/IP washings, and tumor cells collected for research purposes. With your permission we would like to store them after the study ends for future analysis as new things are learned including about the immune system and cancer. Leftover samples may be sent to laboratories outside of the University of Minnesota if specialized testing cannot be performed locally. There is no cost to you or your insurance company for long-term storage. If you agree to storage now and later change your mind, you may contact a member of the research team and request that any remaining identifiable samples be destroyed.

# Use of Identifiable Research Related Samples and/or Health Information

Please indicate whether you will allow the identifiable research related samples and/or health information to be used for future research by putting your initials next to one of the following choices:

| <b>NO</b> , my identifiable research related samples and/or health information |
|---|
| may not be used for future research. They may be used for this study |
| only. |
| <b>YES</b> , my identifiable research related samples and/or health information |
| may be used for other future research studies. |

# **Signature Block:**

| Your signature documents your permission to take with a copy of this signed and dated document. | e part in this research. You will be provided |
|---|---|
| Signature of Participant | Date |
| Printed Name of Participant | |
| Signature of Person Obtaining Consent | <br>Date |

## **STUDY SUMMARY**

## All participants receive:

Printed Name of Person Obtaining Consent

**CY/FLU** - a two day course of outpatient IV (into a vein) chemotherapy with the common anticancer drugs cyclophosphamide (CY) and fludarabine (FLU) or **CY/FLU** for short.

★ FT538 is a NK cell product given after the CY/FLU once a week for 3 weeks in a row as a short infusion through the IP catheter.



## Participants enrolled in Dose Cohort 5 or Dose Cohort 6:

**★ Enoblituzumab** is given as an IV (into a vein) infusion before CY/FLU and approximately 1 week before FT538. Enoblituzumab may continue every 3 weeks until disease progression or unacceptable side effects

#### STUDY TREATMENT PLAN:

This is an early in human study for each of the investigational products (FT538 and enoblituzumab) and a 1<sup>st</sup> in human study for the combination. For this reason, the U.S. Food and Drug Administration (FDA) requires a very careful approach to study treatment. Up to 6 Dose Cohorts will be tested in this study. The dose levels of FT538 match those being tested in other ongoing FT538 studies using intravenous (IV) administration. You will be told which cohort is enrolling when you are told about this study:

| DOSE | STUDY TREATMENT PLAN |
|---|---|
| COHORT | |
| 1 | Low dose of FT538 by IP infusion once a week for 3 weeks |
| 2 | Medium dose of FT538 by IP infusion once a week for 3 weeks |
| 3 | Medium high dose of FT538 by IP infusion once a week for 3 weeks |
| 4 | High dose of FT538 by IP infusion once a week for 3 weeks |
| 5 | Enoblituzumab by IV infusion before CY/FLU and FT538 (at 1 Dose Cohort |
| | drop from the highest Dose Cohort from 1-4) with the option to continue |
| | enoblituzumab every 3 weeks after the FT538 is completed. |
| 6 | Enoblituzumab by IV infusion before CY/FLU and FT538 (at highest Dose |
| | Cohort from 1-4) with the option to continue enoblituzumab every 3 weeks |
| | after the FT538 is completed. |

### **ENROLLMENT PLAN:**

Participants are enrolled and receive the study treatment in this study according to rules for moving from one Dose Cohort to the next.

<u>Start with 1 participant per Dose Cohort</u> until the first unacceptable side effect or Dose Cohort 6 is reached. A minimum of 4 weeks pass from the 1<sup>st</sup> FT538 infusion of a current participant to observe for late side effects and the enrollment of the next participant.

If the 1<sup>st</sup> four Dose Cohorts are completed no unacceptable side effect, the 5<sup>th</sup> participant receives enoblituzumab plus FT538 at one Dose Cohort below the highest level tested (Dose Cohort 3 FT538 dose). Dose Cohort 6 is enoblituzumab plus FT538 at the highest level tested (Dose Cohort 4 FT538 dose).

At the 1<sup>st</sup> unacceptable side effect, the current Dose Cohort is expanded to 3 participants and a minimum of 3 participants are enrolled into all future Dose Cohorts with using a more extensive list of unacceptable side effects. A minimum of 14 days must past between the 1<sup>st</sup> and 2<sup>nd</sup> participant in a Dose Cohort and a new Dose Cohort cannot be assigned until a minimum of 4 weeks pass from the 3rd participant's 1<sup>st</sup> FT538 infusion.

Enrollment continues until 33 participants are treated or 10 participants in a row are treated at the same dose level.